CLINICAL TRIAL: NCT00520897
Title: Effect of Integrase Inhibitor (MK-0518) on Decay of Low Level Viral Replication in HIV Reservoirs in Infected Individuals Who Initiated Conventional Antiretroviral Therapy During the Chronic Phase of Infection
Brief Title: Integrase Inhibitor (MK-0518) Viral Decay
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Immunodeficiency Research Collaborative (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 038-00
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: HIV Infections
Keywords: chronic HIV infection; Human Immunodeficiency Virus; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Raltegravir Potassium; Leukapheresis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- MK0518 + cART (Experimental): Raltegravir + standard of care combined antiretroviral therapy
  Interventions: Drug: Raltegravir (MK0518); Procedure: Leukopheresis; Procedure: Sigmoid Biopsy
- Placebo + cART (Placebo Comparator): Placebo + standard of care combined antiretroviral therapy
  Interventions: Drug: Placebo; Procedure: Leukopheresis; Procedure: Sigmoid Biopsy

INTERVENTIONS:
Drug: Raltegravir (MK0518) — 400mg BID; 48 weeks
  Arms: MK0518 + cART
Drug: Placebo — 400mg QD
  Arms: Placebo + cART
Procedure: Leukopheresis — pack of cells as per protocol
Procedure: Sigmoid Biopsy — gut samples as per protocol

SUMMARY:
The eradication of HIV by antiretroviral therapy has thus far been elusive. It has been consistently demonstrated that a pool of latently infected, resting CD4+ T cells persists in the majority of HIV-infected individuals receiving antiretroviral therapy in whom plasma viremia has been successfully suppressed for prolonged periods of time; this pool has emerged as the major obstacle in achieving the eradication of HIV. We believe that MK-0518 can further the decay and suppression of HIV-1 in patients who have been virologically suppressed for a prolonged period of time on effective cART (≥ 4 years).

DETAILED DESCRIPTION:
The trial is a prospective, double-blind, randomized, placebo-controlled study with two phases: phase I to 48 weeks and phase II to 96 weeks with the primary analysis at 48 weeks. HIV-infected individuals who are taking their first standard cART regimen for at least four years with complete viral suppression. Upon enrollment, he/she will be randomized to one of two arms: the MK-0518 arm or the control arm. As each participant reaches week 48, he/she will be unblinded and those in the MK-0518 arm will continue taking MK-0518. Based on the results of an interim analysis, the control arm will be rolled over to receive MK-0518 for 48 weeks. After the screening, baseline visits and week 4 safety visit, follow-up visits will occur every 8 weeks for both arms.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be HIV-1 infected
2. Participant must be 18 years old
3. Participant must be taking first standard cART with 2-3 NRTIs and 1-2 PIs or an NNRTI for at least four years (first cART regimen may include changes due to toxicity but not due to virologic failure).
4. Participant must have a VL < 50 copies/ml (using the standard available methods of detection) during the entire time on standard cART except for initial fall of VL and a maximum of two non-consecutive blips of < 100 copies/ml that the study investigator deems to be not clinically significant
5. Female participant must agree to use two methods of birth control or abstinence during the period of the study
6. Participant has to have signed full informed consent

Exclusion Criteria:

1. Participant who would have difficulty participating in a trial due to non-adherence or substance abuse
2. Participant who has taken mono or dual antiretroviral therapy in the past
3. Participant who has had a VL > 50 copies/ml on any antiretroviral regimen
4. Participant with any of the following abnormal laboratory test results in screening:

   * Hemoglobin < 100 g/L
   * Neutrophil count < 750 cells/L
   * Platelet count < 50,000 cells/L
   * AST or ALT > 5X the upper limit of normal
   * Creatinine > 250 mol/L
5. Participant with a malignancy
6. Participant with other significant underlying disease (non-HIV) that might impinge upon disease progression or death
7. Participant with an active AIDS-defining illness in the past six months
8. Participant who is pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-04; Primary Completion 2009-02 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
change of proviral HIV-1 DNA in total CD4+ T cells from baseline to week 48 | 48 weeks
  evaluate the change of proviral HIV-1 DNA in total CD4+ T cells from baseline to week 48 in participants randomized to the raltegravir arm (400mg raltegravir) for 48 weeks in addition to their current standard combination antiretroviral regimen versus the control arm, who remained on their current standard combination antiretroviral regimen.

SECONDARY OUTCOMES:
evaluated the effect of raltegravir intensification on blood CD4+ T cell populations | 48 & 96 weeks
  evaluated the effect of raltegravir intensification on blood CD4+ T cell populations. In addition, after treatment-intensification in both groups at week 48, a post-hoc follow-up of all participants was conducted up to week 96 to examine if raltegravir intensification had any long-term effects on proviral HIV DNA and CD4+ T cell populations in the blood and gut.

CONTACTS AND LOCATIONS:
Overall Officials: Mona Loutfy, MD, Principal Investigator — Women's College Hospital
Locations (1):
- Maple Leaf Medical Clinic, Toronto, Ontario, Canada